CLINICAL TRIAL: NCT06074822
Title: Constitution of a Collection of Residues of Neuromuscular Biopsies From Patients Taken as Part of Their Health Care at the Bordeaux University Hospital for Neuromuscular Disease and Use for Research Projects
Brief Title: Research Biobank From Neuromuscular Biopsy Residues (in the Context of Care)
Acronym: COLMYONEU
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/26
Record Dates: First submitted 2023-08-17; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-08

CONDITIONS: Neuromuscular Diseases; Muscle; Nerve
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — collection of remains of neuromuscular biopsy samples (nerve and muscles)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Constitution of biocollection: Collection of remains of neuromuscular biopsy samples (nerve and muscles)
  Interventions: Other: Residual neuromuscular biopsy

INTERVENTIONS:
Other: Residual neuromuscular biopsy — recovery of residual neuromuscular biopsy (nerve ans muscle)

SUMMARY:
Neuromuscular diseases are rare diseases for which significant progress has been made in the context of diagnosis thanks to advances in molecular techniques, but the intimate mechanisms of lesion formation remain poorly understood. Advances in cellular and molecular biology, the development of a few animal models, such as transgenic mice, which make it possible to mimic human pathology have made it possible to better understand the physiopathology of these diseases. However, they still do so very imperfectly and incompletely, making it even more necessary than ever to study diseased human muscle tissue to find new avenues of research or to confirm results obtained by experimentation.

The purpose of this collection of tissue samples for neuro-muscular purposes is to collect such samples under the best conditions in order to promote basic and translational research on muscle diseases.

This is why the CHU de Bordeaux wishes to keep the remainders of samples taken as part of the treatment to constitute a collection of biological samples and associated data kept according to quality standards and in compliance with the regulations in force.

DETAILED DESCRIPTION:
The "COLMYONEU" project is a project to collect leftover frozen neuromuscular biopsy samples from patients taken as part of their health care at the Bordeaux University Hospital for neuromuscular disease.

Its main objective is to store, under the conditions of the CRB standard, residual biological samples from patients with neuromuscular symptoms.

ELIGIBILITY:
Inclusion criteria

* Patients treated at Bordeaux University Hospital (neurology services, neuropediatrics), rheumatology, medical genetics for suspected neuromuscular disease.
* Men and women are affected, adults and minors.

Exclusion criteria

- no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with neuromuscular symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2053-06-25 (Estimated); Study Completion 2053-06-25 (Estimated)

PRIMARY OUTCOMES:
Constitution of a biocollection | 30 years
  Collection of leftover frozen neuromuscular biopsy samples from patients taken as part of their health care at the Bordeaux University Hospital for neuromuscular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Laure NEGRIER, Pr, Principal Investigator — Université Hospital, Bordeaux
Locations (1):
- Université Hospital, Bordeaux, Bordeaux, France